CLINICAL TRIAL: NCT02084030
Title: Screening of Susceptibility Genes in Postoperative Cognitive Dysfunction After On-pump Cardiac Surgery
Brief Title: Screening of Susceptibility Genes in Postoperative Cognitive Dysfunction(POCD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, HailongDong, MD, PhD, Xijing Hospital
Other Study IDs: DONG2014POCD
Record Dates: First submitted 2014-03-04; First posted 2014-03-11 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Cardiac Surgery Patients
Keywords: cardiac surgery; POCD; GWAS; Susceptibility gene

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: blood collected one day before surgery
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Experimental: Patient with POCD: Patients who suffer from POCD after surgery. The mini-mental state examination scale decline more than 1 SD of baseline after surgery.
- Sham Comparator: patient without POCD: Patients who don't suffer from POCD after surgery. There is no obvious difference between pre-operation and post-operation in mini-mental state examination scale

SUMMARY:
The aim of this study is to perform a whole-genome linkage analysis for identification of the susceptibility loci for POCD

DETAILED DESCRIPTION:
BACKGROUND: Postoperative cognitive dysfunction is probably the most frequent type of postoperative cognitive impairment. As it mainly affect the elderly population, POCD is receiving increasing attention. However, the pathophysiology of POCD remains incompletely understood. No study had elucidate why somebody are apt to suffer from POCD, but others not. In current study, we try to use GWAS technology to find out whether there is a correlation between POCD and gene specificity.

DESIGNING: 120 patients will be screened who are schedule to receive selective on-pump cardiac surgery， 5 ml blood of the patient will be collected before anesthesia induction. Investigetors will measure the cognitive function of the patients one day before surgery and 7 d after surgery and identify whether the patient suffer from POCD used in MMSE test. Randomly select 36 patients who suffer from POCD and 36 patients without POCD(control), GWAS technology will be used to screen the susceptibility gene between these two groups.

EXPECTED RESULTS ：Find out some susceptibility genes correlate to POCD.

CONCLUSIONS: The patients who are apt to suffer from POCD have some special susceptibility genes differ from normal people.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 60 to 75 years old;
2. Schedule for on-pump cardiac surgery;
3. undergoing full intravenous anesthesia;
4. without hepatic, renal, pulmonary disease or full intravenous anesthesia surgery history;
5. Gave the informed consent.

Exclusion Criteria:

1. Emergency surgery;
2. A history of cerebrovascular disease;
3. The history of mental disease;
4. Long term use of sedative and antidepressant drugs;
5. Alcoholism;
6. serious vision, hearing impairment and inapprehensive language;
7. chromosomal abnormalities;
8. blood disease;
9. refused to sign the informed consent.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Old patient(>60 y) who are schedule to receive of-pump cardiac surgery.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
single nucleotide polymorphisms(SNPs) of each patient | about 10 minutes before anesthesia induction

SECONDARY OUTCOMES:
mini-mental state examination scale | one day before surgery, 7 d after surgery
  the cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Dong, MD,PhD, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China